CLINICAL TRIAL: NCT05149976
Title: Establishment of Voice Analysis Cohort for Development of Monitoring Technology for Dysphagia
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Other Study IDs: B-2109-707-303
Record Dates: First submitted 2021-11-01; First posted 2021-12-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal group: * A person judged normal among VFSS (video fluoroscopic swallowing study) examiners
  * Normal subjects without symptoms of dysphagia
  Interventions: Diagnostic Test: Voice recording before and after dietary intake
- Residue Group: - As a result of VFSS (video fluoroscopic swallowing study), the subjects who have residues left around the pharynx or airway
  Interventions: Diagnostic Test: Voice recording before and after dietary intake
- Aspiration Group: - VFSS (video fluoroscopic swallowing study) test result, the subjects who have aspiration in the airway
  Interventions: Diagnostic Test: Voice recording before and after dietary intake

INTERVENTIONS:
Diagnostic Test: Voice recording before and after dietary intake — * A person who is scheduled to undergo a VFSS test, and his/her voice is recorded before and after eating for the VFSS test
  * For general subjects, only voice recordings were conducted before and after food/water intake without a VFSS test.

SUMMARY:
Collection of basic data to develop a technique for monitoring the state of dysphagia using voice analysis.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of the patient group

  * Patients scheduled for VFSS examination and normal person (without dysphagia) capable of recording voice (selected as a control group for comparison of voice indicators with patients with dysphagia)
  * Patients who can record voices such as "Ah for 5 seconds", "Ah. Ah. Ah.", "umm~~~"
* Inclusion criteria of the control group: Patients unable to speak, Patients who cannot follow along, If the VFSS test is a retest
* Setting: Hospital rehabilitation department
* Intervention: After obtaining the consent form for the patient scheduled for the VFSS test, "Ah for 5 seconds", after clearing the throat, "Ah for 5 seconds", briefly cut with a high-pitched sound, "Ah. Ah. Ah", close your lips lightly and make a "ummm~~~~" sound, and record 2 times each.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysphagia and scheduled for VFSS testing
* Patients who can record voice such as "Ah for 5 seconds", "Ah. ah. ah", or "Um~~"
* Normal people (without dysphagia symptoms) who can record voice (additionally recruited for comparison of voice indicators with patients with dysphagia)

Exclusion Criteria:

* Patients who cannot speak.
* Patients who cannot speak according to the researcher's instructions.
* Patients whose VFSS test was reexamined

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Normal Group
    1. Among those scheduled for VFSS due to symptoms of dysphagia, patients whose reading result was judged normal
    2. General subjects without signs or symptoms of dysphagia
  * Residue Group
    1) Among those scheduled for VFSS examination due to symptoms of dysphagia, patients who had residues left in the pharynx or airway as a result of reading
  * Aspiration
    1) Among those scheduled for VFSS examination due to symptoms of dysphagia, aspiration occurred in the airway as a result of reading
  * No limiting criteria for age and underlying disease were established in all groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of machine learning prediction model using voice change before and after dietary intake | day 1
  Accuracy measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice changes before and after dietary intake.

SECONDARY OUTCOMES:
mAP (mean Average Precision) of machine learning prediction model using voice change before and after dietary intake | day 1
  mAP measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice changes before and after dietary intake.
Recall of machine learning prediction model using voice change before and after dietary intake. | day 1
  Recall measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice changes before and after dietary intake.
AUC (Area Under the ROC curve) of machine learning prediction model using voice change before and after dietary intake. | day 1
  AUC measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice changes before and after dietary intake.
Accuracy of machine learning prediction model using only voice after dietary intake. | day 1
  Accuracy measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice only voice after dietary intake.
mAP (mean Average Precision) of machine learning prediction model using only voice after dietary intake. | day 1
  mAP measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice only voice after dietary intake.
Recall of machine learning prediction model using only voice after dietary intake. | day 1
  Recall measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice only voice after dietary intake.
AUC (Area Under the ROC curve) of machine learning prediction model using only voice after dietary intake. | day 1
  AUC measures how well machine learning predicts three groups ('Normal', 'Residue', 'Aspiration') according to voice only voice after dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Juseok Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim JM, Kim MS, Choi SY, Lee K, Ryu JS. A deep learning approach to dysphagia-aspiration detecting algorithm through pre- and post-swallowing voice changes. Front Bioeng Biotechnol. 2024 Aug 2;12:1433087. doi: 10.3389/fbioe.2024.1433087. eCollection 2024. PMID 39157445
- [Derived] Kim JM, Kim MS, Choi SY, Ryu JS. Prediction of dysphagia aspiration through machine learning-based analysis of patients' postprandial voices. J Neuroeng Rehabil. 2024 Mar 30;21(1):43. doi: 10.1186/s12984-024-01329-6. PMID 38555417